CLINICAL TRIAL: NCT03289156
Title: Strategies for Responding to Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jolene Jacquart, Graduate Student, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2017-05-0011
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Stress
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arousal Reappraisal (Active Comparator): Brief educational intervention about the stress response and arousal reappraisal
  Interventions: Behavioral: Arousal Reappraisal
- Exercise (Active Comparator): Three 5-minute bouts of aerobic exercise at increasing intensities
  Interventions: Behavioral: Exercise
- Arousal Reappraisal + Exercise (Experimental): Brief educational intervention about the stress response and arousal reappraisal followed by three 5-minute bouts of aerobic exercise at increasing intensities with practice applying the arousal reappraisal learned earlier.
  Interventions: Behavioral: Arousal Reappraisal; Behavioral: Exercise
- Control (No Intervention): Time-matched rest

INTERVENTIONS:
Behavioral: Arousal Reappraisal — Brief readings educating about the stress response and usefulness of arousal reappraisal.
  Arms: Arousal Reappraisal; Arousal Reappraisal + Exercise
Behavioral: Exercise — Three 5-minute bouts of exercise at increasing intensities (65%, 75%, and 85%) with 5-15 minute breaks in-between for recovery.
  Arms: Arousal Reappraisal + Exercise; Exercise

SUMMARY:
The purpose of this study is to examine whether changes in psychological and physiological responses differ based on different strategies for responding to stress.

DETAILED DESCRIPTION:
The purpose of this study is to examine whether changes in psychological and physiological responses differ based on different strategies for responding to stress. Different strategies being examined in this study include exercise and arousal reappraisal.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18 to 35
* Speaks English fluently
* Passes the Physical Activity Readiness Questionnaire-Plus
* Mild to Moderate depression symptoms as measured by the Beck Depression Inventory-II (a score ≥14 but ≤25)

Exclusion Criteria:

* Hearing or visually impaired such that it will interfere with ability to participate effectively
* Currently exercising regularly, defined as exercising at a moderate-intensity more than 2 times a week, for at least 20 minutes each time.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Stress Reappraisal | One day
  Self-report ratings of appraisal of a lab based stressor as threatening or challenging.

SECONDARY OUTCOMES:
Psychological Response to Stress | One day
  Self-report ratings of perceived stress, anxiety, and fear in response to a lab based psychosocial stressor.
Physiological Response to Stress | One day
  Heart rate in response to a lab based psychosocial stressor as threatening or challenging.

CONTACTS AND LOCATIONS:
Overall Officials: Jolene Jacquart, MA, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No